CLINICAL TRIAL: NCT02707796
Title: Evaluation of the Correlation Between Partial Oxygen Pressure and Oxygen Reserve Index, and Sensitivity and Specificity of Oxygen Reserve Index in Patients Undergoing Hemicolectomy
Brief Title: Correlation Between Partial Oxygen Pressure and Oxygen Reserve Index
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr Cigdem Akyol Beyoğlu, MD, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 386986
Record Dates: First submitted 2016-03-02; First posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: COLON CANCER
Keywords: oxygen reserve index, partial oxygen pressure, hemicolectomy
MeSH Terms: conditions — Colonic Neoplasms | interventions — Colectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hemicolectomy (Experimental): Oxygen reserve index and partial oxygen pressure will be noted for patients undergoing hemicolectomy
  Interventions: Procedure: Hemicolectomy

INTERVENTIONS:
Procedure: Hemicolectomy

SUMMARY:
Oxygen reserve index (ORI) measured by multiple wave pulse co-oximeter is a new technological development in medical science. Our aim in this study is to identify the correlation between arterial oxygen pressure (PaO2) and ORI, and to identify the specificity and sensitivity of ORI as a tool to prevent hypoxia and hyperoxia in abdominal surgery patients.

DETAILED DESCRIPTION:
Patients aged between 20-55 years old,American Society of Anesthesiologists physical status 1-2 who will have hemicolectomy will be included to the study. If hemodynamic instability or a sudden decrease in oxygen saturation by pulse oximetry (SpO2) occurs, arterial blood gas analysis will be taken from the patient and ORI, SpO2, PaO2, and arterial oxygen saturation (SaO2) will be recorded. The primer endpoint of the study is to identify the correlation between PaO2 and ORI, seconder end-point is to identify the specificity and sensitivity of ORI as a detector of PaO2. Pearson test for correlation, regression analysis for sensitivity and specificity will be performed. The study will include 240 patients according to power analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 20-55 years old
* American Society of Anesthesiologists physical status I-II
* Patients undergoing hemicolectomy

Exclusion Criteria:

* Chronic obstructive and restrictive pulmonary disease
* Diabetes Mellitus
* Ischemic heart disease
* Peripheric artery disease.
* Operations longer than 200 minutes, requirement transfusion of more than 1 U erythrocyte suspension, and requirement of vasopressor or inotrope infusion will be excluded from the study

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the correlation between partial oxygen pressure in arterial blood sample and oxygen reserve index calculated by pulse co-oximetry, and sensitivity and specificity of oxygen reserve index in patients undergoing hemicolectomy | oxygen reserve index and peripheric oxygen saturation will be recorded before and after induction of anesthesia, and every 5 minutes and arterial partial oxygen pressure in every 30 minutes during hemicolectomy.

SECONDARY OUTCOMES:
Sensitivity and specificity of oxygen reserve index | During Hemicolectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Cigdem Akyol Beyoglu, Istanbul, Turkey (Türkiye)